CLINICAL TRIAL: NCT07275463
Title: SPECT/CT Imaging of Gastrin-releasing Peptide Receptor Expression in Breast Cancer With Different Estrogen Receptor Expression Using Technetium-99m-labelled DB8 [99mTc]Tc-DB8
Brief Title: [99mTc]Tc-DB8 Accumulation in Primary Tumor in Breast Cancer With Positive and Negative Estrogen Receptor Expression
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Molecular imaging of GRPR
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Primary Breast Cancer
Keywords: [99mTc]Tc-DB8; Breast Cancer; Gastrin-releasing peptide receptor expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Diagnostic SPECT for GRPR expression in primary tumour
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast cancer patients with positive estrogen receptor expression (Experimental): Assessment of [99mTc]Tc-DB8 accumulation in primary tumour of breast cancer patients with positive estrogen receptor expression.
  Interventions: Drug: [99mTc]Tc-DB8
- Breast cancer patients with negative estrogen receptor expression (Experimental): Assessment of [99mTc]Tc-DB8 accumulation in primary tumour of breast cancer patients with negative estrogen receptor expression.
  Interventions: Drug: [99mTc]Tc-DB8

INTERVENTIONS:
Drug: [99mTc]Tc-DB8 — One single injection of [99mTc]Tc-DB8, followed by SPECT/CT imaging 2 hours after the injection
  Other Names: Technetium-99m-labelled DB8

SUMMARY:
The study should evaluate the [99mTc]Tc-DB8 accumulation in primary tumour of breast cancer patients with positive and negative estrogen receptor expression.

DETAILED DESCRIPTION:
The aim of the study is to determine gastrin-releasing peptide receptor expression in primary breast cancer patients with positive and negative estrogen receptor expression before any systemic or local treatment.

Phase II. Assessment of [99mTc]Tc-DB8 accumulation in primary tumors with positive and negative estrogen receptor expression in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Availability of results from estrogen receptor status by Immunohistochemistry previously determined on material from the primary tumor
3. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 109/L
   * Hemoglobin: > 80 g/L
   * Platelets: > 50.0 x 109/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
4. A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
5. Subject is capable to undergo the diagnostic investigations to be performed in the study
6. Informed consent

Exclusion Criteria:

1. Any system therapy (chemo-/targeted therapy)
2. Second, non-breast malignancy
3. Active current autoimmune disease or history of autoimmune disease
4. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
[99mTc]Tc-DB8 uptake in primary breast tumor | 2 hours
  SPECT/СT-based [99mTc]Tc-DB8 uptake in primary breast tumor with positive and negative estrogen receptor expression (SUVmax)
[99mTc]Tc-DB8 background uptake value | 2 hours
  SPECT/CT-based [99mTc]Tc-DB8 background uptake value (SUVmax)
Tumor-to-background ratio (SPECT/CT) | 2 hours
  The SPECT/CT-based tumor-to-background ratio will be calculated as follows: the value of [99mTc]Tc-DB8 uptake coinciding with tumor lesions (counts) will be divided by the value of [99mTc]Tc-DB8 uptake coinciding with the regions without pathological findings (SUVmax)

SECONDARY OUTCOMES:
Estrogen receptor positive vs estrogen receptor negative [99mTc]Tc-DB8 uptake | 2 hours
  To evaluate the threshold values of [99mTc]Tc-DB8 accumulation for differentiation of estrogen receptor status in primary tumors in breast cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, Prof, Principal Investigator — Tomsk NRMC
Locations (1):
- Russia Tomsk NRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.